CLINICAL TRIAL: NCT00653419
Title: Comparative, Randomized, Single-Dose, 2-Way Crossover Bioavailability Study of Par and Bristol-Myers Squibb (Buspar) 15 mg Buspirone HCl Tablets in Healthy Adult Males Under Fasting Conditions Following Administration of a 30 mg Dose
Brief Title: Bioavailability Study of (Buspar) Buspirone HCl Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Phoenix International Life Sciences, Inc. (Industry)
Responsible Party: Alfred Elvin/Director of Biopharmaceutics, Par Pharmaceutical Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 980563
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: To Determine Bioequivalence Under Fasting Conditions
Keywords: bioequivalence; buspirone HCl; fasting
MeSH Terms: conditions — Fasting | interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received the Par formulated product (Buspirone HCl) under fasting conditions
  Interventions: Drug: buspirone HCl
- B (Active Comparator): Subjects received the Bristol-Myers Squibb formulated product (Buspar) under fasting conditions
  Interventions: Drug: Buspar

INTERVENTIONS:
Drug: buspirone HCl — Tablets, 30 mg, single-dose
  Other Names: Buspar
  Arms: A
Drug: Buspar — Tablets, 30 mg, single-dose
  Other Names: buspirone HCl
  Arms: B

SUMMARY:
To compare the single-dose bioavailability of Par and Bristol-Myers Squibb Buspirone HCl Tablets

DETAILED DESCRIPTION:
To compare the single-dose bioavailability of Par and Bristol-Myers Squibb (Buspar) 15 mg Buspirone HCl Tablets under fasting conditions, following administration of a 30 mg dose

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 18-45 years of age
* Weighing at least 60 kg, who are within 10% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983)
* Physical examination and laboratory tests of hematologic, hepatic and renal functions
* Medically healthy subjects with clinically normal laboratory profiles will be enrolled in the study

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease
* The presence of alcoholism or drug abuse within the past year
* Hypersensitivity or idiosyncratic reaction to buspirone HCl
* Subjects who have been receiving monoamine oxidase inhibitors
* Subjects who have been on an abnormal diet (for whatever reason) during the 28 days preceding the study
* Subjects who, through completion of the study, would have donated in excess of 500 mL blood in 14 days, or 500-750 mL of blood in 14 days (unless approved by Principal Investigator, 1000 mL blood in 90 days, 1250 mL blood in 120 days, 1500 mL blood in 180 days, 2000 mL blood in 270 days, 2500 mL blood in 1 year
* Subjects who have participated in another clinical trial within 28 days of study start

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 1998-06; Primary Completion 1998-09 (Actual); Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Serfaty, MD, Principal Investigator — Phoenix International Life Sciences, Inc.
Locations (1):
- Phoenix International Life Sciences, Inc., Saint-Laurent, Quebec, Canada